CLINICAL TRIAL: NCT05868096
Title: Improving Occupational Therapy Students' Holistic Care Competencies Through a Structured Holistic Thinking Curriculum: a Mixed Design
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N202212038
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-07

CONDITIONS: Holistic Care Competencies of Occupational Therapy Students
Keywords: Holistic health care; occupational therapy student; mind map

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): During the 12 weeks of the internship, the experimental group took a pre-test after a case report-1 in weeks 4-5, which included completing the holistic thinking case analysis form and the personal learning self-efficacy questionnaire, followed by a 2-hour structured holistic thinking course. At the end of the session, subjects took the first post-test, revised the case analysis form completed in the pre-test based on the case report-1 observed in the pre-test, and completed the personal learning self-efficacy questionnaire and the satisfaction questionnaire again. During weeks 6-11 of the internship, participants continue to receive clinical practice training in assessment, intervention planning, and patient intervention skills. In weeks 11-12 of the internship, subjects took a second post-test after reading case report-2, which included completing the holistic thinking case analysis form and again completing the personal learning self-efficacy questionnaire.
  Interventions: Other: Structured holistic thinking course(2 hr)
- Control group (Active Comparator): During the 12 weeks of the internship, the control group had no structured holistic thinking course. During weeks 4-5 of the internship, after viewing case report-1, a pretest consisting of completing the holistic thinking case analysis form and the personal learning self-efficacy questionnaire was completed and a holistic thinking case analysis form - introductory version was given. Subjects will revise the holistic thinking case analysis form completed in the pretest and complete the personal learning self-efficacy questionnaire again. During weeks 6-11 of the internship, participants continue to receive clinical practice training in assessment, intervention planning, and patient intervention skills. In weeks 11-12 of the internship, subjects received the post-test, viewed the case report-2, and were given the holistic thinking case analysis form - introductory version and completed the holistic thinking case analysis form and the personal learning self-efficacy questionnaire.
  Interventions: Other: Clinical practice training

INTERVENTIONS:
Other: Structured holistic thinking course(2 hr) — The holistic thinking curriculum was designed as a structured program using mind maps, case-based discussions, and clinical observations to integrate physical, psychological, social, and spiritual aspects.
  Arms: Experimental group
Other: Clinical practice training — there is no holistic thinking curriculum.Using the holistic thinking case study form - introductory version self-study
  Arms: Control group

SUMMARY:
Background: Occupational therapy emphasizes the holistic approach, but occupational therapy students are unable to use holistic thinking to design holistic solutions for cases immediately during their internship due to their lack of clinical experience, which requires extensive guidance from clinical occupational therapist.

Study Aim: To improve the holistic care competencies of occupational therapy students using a structured holistic thinking curriculum.

Methods: The study population was occupational therapy interns from a northern teaching hospital. The holistic thinking curriculum was designed as a structured program using mind maps, case-based discussions, and clinical observations to integrate physical, psychological, social, and spiritual aspects. The experimental group took a pre-test after a case report in weeks 4 and 5, a first post-test and course satisfaction after the first structured holistic thinking course, and a second structured holistic thinking course with a second post-test and course satisfaction in weeks 11 and 12; the control group had no course but had a guided version of the holistic thinking case study form for independent study, and the control and experimental groups were tested pre and post using the holistic thinking case study form and the personal learning self-efficacy scale.

Data analysis: Quantitative data for the holistic thinking case study form were determined by three occupational therapists with at least 5 years of teaching experience through consensus conferences to determine the degree of compliance of the case study form with holistic care, and differences between the holistic thinking case study form and the personal learning self-efficacy scale were determined by Kruskal-Wallis with a p-value of 0.05. Qualitative data for the holistic thinking case study form were determined by three occupational therapists with at least 5 years of teaching experience to determine the degree of compliance of the case study form with holistic care and regular meetings were held to achieve consistency in coding.

ELIGIBILITY:
Inclusion Criteria:

1. occupational therapy students who were interns at the Shuanghe Hospital, Ministry of Health and Welfare
2. students who could read, write, and communicate in Chinese
3. students who were 20 years of age or older.

Exclusion Criteria:

1. those who could not attend the entire course
2. those who could not complete the 12-week internship.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The quantitative data of the Holistic Thinking Case Analysis Form | Change from baseline after immediate intervention/Change from baseline at week 12
  The Holistic Thinking Case Analysis Form: Taken from cases (caregivers) to see if subjects can analyze holistic abilities/problems based on physical, mental, social and spiritual aspects. Higher scores indicate better analysis of the problem and are quantitative data. The holistic occupational therapy intervention plan extract looks at whether the subject can present an occupational therapy intervention plan with the concept of holistic care, which is qualitative. The higher the score, the more appropriate it is, which is quantitative data. The above information was coded and analyzed by three occupational therapists with more than five years of teaching experience, and quantitative information was determined through consensus conferences.
MSLQ:Motivated Strategies for Learning Questionnaire | Change from baseline after immediate intervention/Change from baseline at week 12
  Measuring subjects' learning self-efficacy

SECONDARY OUTCOMES:
Course Satisfaction Questionnaire | After each training session(week 4-5/week 11-12)
  The purpose of the questionnaire was to understand the subjects' satisfaction, usefulness, and suggestions regarding the course content and to increase the subjects' connection to the holistic care curriculum, clinical experience, and skills knowledge through course reflection.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Profetto-McGrath J. Critical thinking and evidence-based practice. J Prof Nurs. 2005 Nov-Dec;21(6):364-71. doi: 10.1016/j.profnurs.2005.10.002. PMID 16311232
- [Background] Girot EA. Graduate nurses: critical thinkers or better decision makers? J Adv Nurs. 2000 Feb;31(2):288-97. doi: 10.1046/j.1365-2648.2000.01298.x. PMID 10672085
- [Background] Holden RJ. Lean Thinking in emergency departments: a critical review. Ann Emerg Med. 2011 Mar;57(3):265-78. doi: 10.1016/j.annemergmed.2010.08.001. Epub 2010 Oct 29. PMID 21035904
- [Background] McCombie RP, Antanavage ME. Transitioning From Occupational Therapy Student To Practicing Occupational Therapist: First Year of Employment. Occup Ther Health Care. 2017 Apr;31(2):126-142. doi: 10.1080/07380577.2017.1307480. Epub 2017 Apr 24. PMID 28436709
- [Result] Chen SL, Liang T, Lee ML, Liao IC. Effects of concept map teaching on students' critical thinking and approach to learning and studying. J Nurs Educ. 2011 Aug;50(8):466-9. doi: 10.3928/01484834-20110415-06. Epub 2011 Apr 15. PMID 21524017
- [Result] D'Antoni AV, Zipp GP, Olson VG, Cahill TF. Does the mind map learning strategy facilitate information retrieval and critical thinking in medical students? BMC Med Educ. 2010 Sep 16;10:61. doi: 10.1186/1472-6920-10-61. PMID 20846442
- [Result] Jenicek M, Croskerry P, Hitchcock DL. Evidence and its uses in health care and research: the role of critical thinking. Med Sci Monit. 2011 Jan;17(1):RA12-7. doi: 10.12659/msm.881321. PMID 21169920
- [Result] Wu HZ, Wu QT. Impact of mind mapping on the critical thinking ability of clinical nursing students and teaching application. J Int Med Res. 2020 Mar;48(3):300060519893225. doi: 10.1177/0300060519893225. PMID 32212879